CLINICAL TRIAL: NCT00168090
Title: Study of Safety and Efficacy of Antihemophilic Factor/Von Willebrand Factor Complex (Humate-P®) Using Individualized Dosing in Pediatric and Adult Surgical Subjects With Von Willebrand's Disease.
Brief Title: Study of Safety and Efficacy of Antihemophilic Factor/Von Willebrand Factor Complex in Surgical Subjects With Von Willebrand Disease (vWD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP7000/1-4002
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Von Willebrand Disease; Blood Coagulation Disorders; Blood Platelet Disorders; Hematologic Disease
Keywords: von Willebrand Factor; Blood Coagulation Disorders; Factor VIII
MeSH Terms: conditions — von Willebrand Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Hematologic Diseases; Hemophilia A | interventions — Factor VIII

INTERVENTIONS:
Drug: Blood coagulation Factor VIII and vWF, human

SUMMARY:
The purpose of this study is to test the safety and effectiveness of Humate-P® to prevent bleeding in patients with von Willebrand Disease who are undergoing surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects of any age
* Clinical and laboratory diagnosis of vWD that can be expected to show no hemostatic response to DDAVP
* Require substitution with vWF/FVIII complex due to a surgery

Key Exclusion Criteria:

* Known significant hemostatic disorder other than vWD
* Acquired vWD
* Known antibodies to FVIII or vWF
* Known platelet type vWD
* Emergency surgery or any surgery with a degree of urgency not permitting completion of a pharmacokinetic assessment required by the study protocol
* History of allergic reaction to Humate-P®
* Treatment with any other investigational drug in the last four weeks before the entry into the study (with exception of trials concerning anti-HIV agents)
* Progressive fatal disease/life expectancy of less than 6 months
* Treatment with DDAVP, cryoprecipitate, whole blood, plasma and plasma derivatives containing substantial quantities of FVIII and/or vWF within 5 days of the pre-surgical pharmacokinetic assessment
* Pediatric patients of insufficient body weight to permit PK sampling
* Woman in the first 20 weeks of pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2001-10; Study Completion 2006-05

PRIMARY OUTCOMES:
To demonstrate the efficacy and safety of HumateP® in preventing excessive bleeding in pediatric and adult surgical subjects with vWD using individualized dosing based on VWF:RCo and FVIII:C monitoring.

SECONDARY OUTCOMES:
To document the pharmacokinetics of Humate-P® in pediatric and adult subjects with various types of vWD.

CONTACTS AND LOCATIONS:
Overall Officials: Marylin J. Manco-Johnson, M.D., Principal Investigator — Mountain States Regional Hemophilia Center, Aurora, Columbia, U.S.
Locations (1):
- Milwaukee, Wisconsin, United States

REFERENCES:
- See also: Click here for more information about this study. — http://allaboutbleeding.com